CLINICAL TRIAL: NCT03732053
Title: The Effectiveness of Physical Rehabilitation in the Enhancement of Proprioceptive and Cognitive Aspects on Alzheimer Disease Patients
Brief Title: The Effectiveness of Global Postural Reeducation on Alzheimer Disease Patients
Acronym: GPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Jasemin Todri, PhD Candidate in Health Science, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BJ8674287
Record Dates: First submitted 2018-04-17; First posted 2018-11-06 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Alzheimer's Type Dementia; Cognitive Decline; Postural; Strain
MeSH Terms: conditions — Cognitive Dysfunction; Sprains and Strains

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPR Intervention Research group (Experimental): A total of 135 subjects with AD in the mild or moderate phase participated in the study from which 90 pertain to research group.The intervention implemented to the patients with AD was the Global Postural therapy which lasted about 30-40 min in repeated sessions of 2 meetings per week by making 48 sessions in total during a six month period.
  Interventions: Other: GPR Intervention Research group
- Control Group (No Intervention): 45 subjects of the study belongs to the control group which has not received the same treatment .

INTERVENTIONS:
Other: GPR Intervention Research group — The research intervention consisted in the reappointment of three GPR therapeutic postures.
  Arms: GPR Intervention Research group

SUMMARY:
This research study is developed on an experimental design with randomized controlled intervention were participated 135 subjects with AD including 45 of the control group. It lasted 6 months with pre-post tests (T0-T1) executed before and after six months of treatment. By having in focus the evaluation of GPR therapy effects on cognitive, proprioceptive, depressive, autonomy, gait and life quality of the above mentioned subjects.

DETAILED DESCRIPTION:
In order to assess the cognitive abilities of the patients a cognitive test was administered which acts through a scale concerning depression and mood evaluation as well as a questionnaire was developed aiming to evaluate the examined subjects' functional abilities: Mini Mental State Examination (MMSE), Quality of Life in Alzheimer Disease (QoL-AD), geriatric Depression Scale (GDS), Barthel Index (BI), Neuropsychiatric Inventory (NPI), Tinetti Scale (TS).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's Disease
* Older than 40 years of age
* Male and female
* Intellectual disability
* Cognitive impairment
* Able to do daily activities on his own
* No presence of any other neurological and psychological disease
* No presence of brain tumors

Exclusion Criteria:

* No presence of Alzheimer's Disease
* Under 40 years old
* Presence of brain tumors
* Neurological patients
* Presence of psychiatric disease
* Depression symptoms
* Presence of neuromuscular disease
* Ictus
* Aggressive patients

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Cognitive Abilities Measurement | Change from baseline cognitive evaluation at 6'th month
  The therapeutist provides the Mini Mental State Examination (MMSE) scale records. The evaluation consits in a 0-30 points-scale. Lower scores imply the severity of dementia.

SECONDARY OUTCOMES:
Quality of Life in Alzheimer's disease (QoL-AD) Questionnaire | Change from baseline cognitive evaluation at 6'th month
  The therapeutist measures in the begining and in the end of the study the quality of life in patients with Alzheimer's disease (QoL-AD). This questionnaire consists in 13 elements referring to the perception that patients have concerning various aspects of their life: mood, health, cognition, environment and functional capacity. The range of scores is 13-52, were higher scores indicate a better life quality.
Geriatric Depression Scale (GDS) Questionnaire | Change from baseline cognitive evaluation at 6'th month
  The version of 15 articles was used, which given its length can be validly and reliably resolved by patients themselves in the quality of a self-report questionnaire aiming to investigate the possible presence of depressive symptoms.
Barthel Index (BI) | Change from baseline cognitive evaluation at 6'th month
  This scale is used by therapist to measure the performance in the basic activities of daily life of AD patients. The maximum score used is 100 points and refers to the patient's independence in all basic daily living activities.
Neuropsychiatric Inventory (NPI) | Change from baseline cognitive evaluation at 6'th month
  This test includes 12 symptoms scored according to the phenomenon severity and frequency. It is a helpful instrument for the therapist because of specifically designed for the assessment of psycho-behavioral disorders in individuals with cognitive impairment.
Tinetti Scale (TS) | Change from baseline cognitive evaluation at 6'th month
  The therapist used the equilibrium sub-scale, which consists in 7 elements and has a score between 0 and 13. Highest scores indicate a better balance.

IPD SHARING:
Plan to Share IPD: No
All participants signed the informed consent and their family members were also informed concerning the purpose of the study. Correspondingly the data were provided by the physiotherapists who performed the above mentioned technique. Thereafter the study was validated and approved by the Ethics Committee of Catholic University of Murcia.

REFERENCES:
- [Derived] Todri J, Lena O, Todri A, Fuentes JM. Does the Global Postural Re-Education Affect the Psychological and Postural Aspects of Alzheimer Disease Patients? A Six Months Quasi-Experimental Study. Curr Alzheimer Res. 2021;18(13):1057-1065. doi: 10.2174/1567205019666211223094811. PMID 34951386